CLINICAL TRIAL: NCT00824538
Title: Pilot Study to Evaluate the Effect of Sunitinib on Occult Tumor Cells in the Bone Marrow of Patients With High Risk Early Stage Breast Cancer
Brief Title: Sunitinib in Treating Patients With Stage I, Stage II, or Stage III Breast Cancer Who Have Tumor Cells in the Bone Marrow
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed prematurely due to emerging data on toxicity and competing trials.
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 077539; 077539 (Other: University of California, San Francisco)
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Results first posted 2014-05-08 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-03

CONDITIONS: Breast Cancer
Keywords: stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Sunitinib; Flow Cytometry; Immunohistochemistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sunitinib (Experimental): Study to evaluate the effect of sunitinib (37.5 mg/day orally for 6 months) on occult tumor cells in the bone marrow of patients with high risk early stage breast cancer
  Interventions: Drug: sunitinib malate; Other: flow cytometry; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: sunitinib malate
Other: flow cytometry
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Sunitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying how well sunitinib works in treating patients with stage I, stage II, or stage III breast cancer who have tumor cells in the bone marrow.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the effect of sunitinib malate on occult tumor cells (OTC) in the bone marrow of patients with high-risk stage I-III breast cancer.

Secondary

* To evaluate the number of patients who are able to tolerate this drug for 6 months and complete the study.
* To evaluate the toxicities of this drug in these patients.
* To evaluate the effects of this drug on OTC in peripheral blood.
* To evaluate correlative markers, including endothelial cells, soluble cKIT, and VEGF.
* To evaluate relapse-free and overall survival of patients treated with this drug.

OUTLINE: Patients receive oral sunitinib malate once daily for 6 months in the absence of disease progression or unacceptable toxicity.

Patients undergo bone marrow aspiration and peripheral blood sample collection at baseline and at 6 and 12 months. Bone marrow aspirate samples are analyzed by IHC and flow cytometry. Peripheral blood samples are analyzed for circulating tumor cells.

After completion of study treatment, patients are followed at 1 and 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed high-risk breast cancer

  * Stage I-III disease
* Has undergone definitive surgery with or without radiotherapy

  * Completely resected disease
* Bone marrow aspirate positive for occult tumor cells, defined as ≥ 10 occult tumor cells/mL by IHC and flow cytometry

  * If the patient received either no adjuvant therapy or hormonal therapy alone, the aspiration may have been performed at diagnosis as part of the large micrometastasis study at UCSF, or following diagnosis if the patient underwent initial surgery elsewhere (or underwent surgery following neoadjuvant therapy for breast cancer)
  * If the patient received adjuvant chemotherapy, the aspiration must have been performed ≥ 3 weeks after completion of chemotherapy
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* ECOG performance status 0-1
* WBC count normal (3.4-10 x 10^9/L)
* Hemoglobin > 9.0 g/dL
* Platelet count normal (140-450 x 10^9/L)
* ANC normal (1.8-6.8 x 10^9/L)
* Serum creatinine ≤ 1.5 times upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 times ULN
* Alkaline phosphatase ≤ 1.5 times ULN
* AST and ALT ≤ 2.5 times ULN
* TSH and T4 levels normal
* LVEF > 50%
* Systolic BP < 140 mm Hg and diastolic BP < 90 mm Hg
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of HIV infection
* No concurrent severe illness that would likely preclude study compliance
* No other malignancy within the past 5 years except basal cell carcinoma of the skin

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior sunitinib malate
* Prior adjuvant chemotherapy, including trastuzumab (Herceptin®), allowed provided it was completed within the past 6 months
* Prior surgery following neoadjuvant chemotherapy or hormonal therapy allowed
* No concurrent potent CYP3A4 inducers
* No concurrent trastuzumab
* Concurrent hormonal therapy or radiotherapy allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-02; Primary Completion 2010-11-10 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hope S. Rugo, MD, Principal Investigator — University of California, San Francisco

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients (pts) were enrolled in this study over the course of a year, from May 2009 through May 2010. A total of 21 patients were screened, and 13 patients, demonstrating ≥ 10 DTCs/mL via bone marrow aspiration, were deemed eligible.
Pre-assignment Details: 13 patients were enrolled, and 11 received 6-month bone marrow aspirations after completing sunitinib treatment.
Groups:
- Sunitinib (SU): Eligible pts were treated with SU for 6 months (mo) at 37.5 mg/day. Concomitant hormonal therapy was allowed. Repeat BM aspirations were performed at 6 mo and one year. DTCs were detected by immunomagnetic enrichment + flow cytometry (IE/FC)
Period: Overall Study
Arm/Group | Sunitinib (SU)
Started | 13 (13 patients entered the study)
Completed | 11
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Sunitinib (SU)
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Disseminated Tumor Cells (DTC) in Bone Marrow
Description: DTCs were detected by immunomagnetic enrichment and flow cytometry (IE/FC) and measured in cells/mL
Time Frame: Baseline, 6 months after start of treatment
Measure: Mean (Full Range); unit: percentage of change
Arm/Group | Sunitinib (SU)
Number analyzed (Participants) | 11
percentage of change | 39 [1 to 90]

2. Secondary Outcome: Number of Patients Who Are Able to Tolerate Sunitinib Malate for 6 Months and Complete the Study
Time Frame: after 6 months from start of treatment
Measure: Number; unit: participants
Groups:
- Sunitinib: Eligible pts were treated with SU for 6 months (mo) at 37.5 mg/day. Concomitant hormonal therapy was allowed. Repeat BM aspirations were performed at 6 mo and one year. DTCs were detected by immunomagnetic enrichment + flow cytometry (IE/FC)
Arm/Group | Sunitinib
Number analyzed (Participants) | 13
participants | 11

3. Secondary Outcome: Participants Affected by Toxicities as Assessed by NCI CTCAE v3.0
Time Frame: up to 7 months after start of treatment
Measure: Number; unit: participants
Arm/Group | Sunitinib (SU)
Number analyzed (Participants) | 13
participants | 13

4. Secondary Outcome: Relapse-free and Overall Survival
Description: Data was not collected due to emerging data on toxicity and competing trials.
Time Frame: up to 3 years from beginning of treatment
Arm/Group | Sunitinib (SU)
Number analyzed (Participants) | 0

5. Secondary Outcome: Effect of Sunitinib Malate on OTC in Peripheral Blood
Description: Data was not collected due to emerging data on toxicity and competing trials.
Time Frame: After one year of treatment
Arm/Group | Sunitinib (SU)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Sunitinib (SU)
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 13/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (SU) (N=13)
ache in the axillary (Reproductive system and breast disorders) | 1
agitation (Psychiatric disorders) | 1
alanine aminotransferase increased (Investigations) | 1
alkaline phosphatase increased (Investigations) | 2
alopecia (Skin and subcutaneous tissue disorders) | 1
anemia (Blood and lymphatic system disorders) | 3
anorexia (Metabolism and nutrition disorders) | 1
anxiety (Psychiatric disorders) | 3
arthralgia (Musculoskeletal and connective tissue disorders) | 8
aspartate aminotransferase increased (Investigations) | 4
back pain (Musculoskeletal and connective tissue disorders) | 2
blood bilirubin increased (Investigations) | 1
Blurred vision (Eye disorders) | 2
bone pain (Musculoskeletal and connective tissue disorders) | 1
breast pain (Reproductive system and breast disorders) | 1
bruising (Injury, poisoning and procedural complications) | 3
chills (General disorders) | 1
congestion (Respiratory, thoracic and mediastinal disorders) | 4
constipation (Gastrointestinal disorders) | 4
cough (Respiratory, thoracic and mediastinal disorders) | 4
creatinine increased (Investigations) | 2
depression (Psychiatric disorders) | 1
diarrhea (Gastrointestinal disorders) | 7
dizziness (Nervous system disorders) | 3
dry eye (Eye disorders) | 2
dry skin (Skin and subcutaneous tissue disorders) | 5
dry throat (Respiratory, thoracic and mediastinal disorders) | 1
dysgeusia (Nervous system disorders) | 2
dyspepsia (Gastrointestinal disorders) | 3
dysphagia (Gastrointestinal disorders) | 1
dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
ears plugged (Ear and labyrinth disorders) | 1
edema face (General disorders) | 1
fatigue (General disorders) | 11
feet numbness (Nervous system disorders) | 1
flashing light (Eye disorders) | 3
flatulence (Gastrointestinal disorders) | 1
floaters (Eye disorders) | 1
hand-foot syndrome (Skin and subcutaneous tissue disorders) | 4
headache (Nervous system disorders) | 7
hip pain (Musculoskeletal and connective tissue disorders) | 2
hot flashes (Vascular disorders) | 4
hyperkalemia (Metabolism and nutrition disorders) | 1
hypernatremia (Metabolism and nutrition disorders) | 1
hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
hypertension (Vascular disorders) | 3
hypoalbuminemia (Metabolism and nutrition disorders) | 1
hypocalcemia (Metabolism and nutrition disorders) | 3
hypokalemia (Metabolism and nutrition disorders) | 2
hypophosphatemia (Metabolism and nutrition disorders) | 1
hypothyroidism (Endocrine disorders) | 4
insomnia (Psychiatric disorders) | 4
lightheadedness (Nervous system disorders) | 1
lumpy breast (Reproductive system and breast disorders) | 1
lymphocyte count decreased (Investigations) | 2
memory impairment (Nervous system disorders) | 1
mucositis oral (Gastrointestinal disorders) | 7
myalgia (Musculoskeletal and connective tissue disorders) | 3
nausea (Gastrointestinal disorders) | 6
neck pain (Musculoskeletal and connective tissue disorders) | 1
neuralgia (Nervous system disorders) | 1
neutrophil count decreased (Investigations) | 12
night sweat (Vascular disorders) | 1
non-cardiac chest pain (General disorders) | 1
numbness in the axillary (Reproductive system and breast disorders) | 1
oral dysesthesia (Gastrointestinal disorders) | 3
pain in extremity (Musculoskeletal and connective tissue disorders) | 12
pain of skin (Skin and subcutaneous tissue disorders) | 1
peripheral sensory neuropathy (Nervous system disorders) | 6
photophobia (Eye disorders) | 1
platelet count decreased (Investigations) | 7
rash (Skin and subcutaneous tissue disorders) | 5
rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
sore throat (Respiratory, thoracic and mediastinal disorders) | 3
subconjunctival hemorrhage (Eye disorders) | 1
urinary frequency (Renal and urinary disorders) | 2
urinary tract infection (Renal and urinary disorders) | 1
vaginal dryness (Reproductive system and breast disorders) | 2
vomiting (Gastrointestinal disorders) | 2
weight loss (Investigations) | 1
white blood cell decreased (Investigations) | 11
white hair (Skin and subcutaneous tissue disorders) | 3
wound infection (Infections and infestations) | 1

LIMITATIONS AND CAVEATS:
The study closed early due to results released from a phase III metastatic breast cancer (MBC) study that demonstrated significant sunitinib toxicity without commensurate clinical benefit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No